CLINICAL TRIAL: NCT00364520
Title: Molecular Epidemiology of Benzene-exposed Workers in Shanghai,China
Brief Title: Molecular Epidemiology of Benzene-exposed Workers.
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Fudan University (Other); University of Cincinnati (Other); ExxonMobil Biomedical Sciences, Inc. (Industry); British Petroleum P.L.C. (Industry); Chevron Corporation (Industry); ConocoPhillips (Industry); Exxon Mobil (Industry); Marathon Ashland (Unknown); Shell Chemicals (Industry)
Responsible Party: Sponsor
Other Study IDs: 02-0037
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Hematologic Diseases
Keywords: Hematologic Diseases; Benzene; Genetic Polymorphisms
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Shanghai Workers: Shanghai Workers
  Interventions: Other: Shanghai workers

INTERVENTIONS:
Other: Shanghai workers

SUMMARY:
The purpose of this study is to investigate the health effects of benzene exposure in workers in Shanghai, China.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the dose-response relationship between benzene exposure and blood diseases in Shanghai workers and to characterize genetic polymorphisms that are associated with increased risk of developing benzene hematotoxicity.

ELIGIBILITY:
Inclusion Criteria:

Worked for at least one year in a monitored environment Have at least one physical examination recorded

-

Exclusion Criteria:

History of cancer, radiation exposure, chemotherapy

-

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Shanghai Workers
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2003-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Investigate the dose-response relationship between benzene exposure and blood diseases in Shanghai workers. | August 2003 - December 2009
  Investigate the dose-response relationship between benzene exposure and blood diseases in Shanghai workers

SECONDARY OUTCOMES:
Characterize genetic polymorphisms that are associated with increased risk of developing benzene hematotoxicity. | August 2003 - December 2009
  Characterize genetic polymorphisms that are associated with increased risk of developing benzene hematotoxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Irons, PhD, Principal Investigator — University of Colorado at Denver and Health Sciences Ctr
Locations (1):
- Joint Sino-US Clinical and Molecular Laboratory (JCML), Shanghai, China